CLINICAL TRIAL: NCT04969003
Title: Reducing Transphobia Among Adolescents Through a Brief Video Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000028980_a
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Transgenderism; Depression
MeSH Terms: conditions — Transsexualism; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transgender male (TM) (Active Comparator): ~90-second video of depressed transgender male
  Interventions: Behavioral: Short videos
- Cis-gender male (CM) (Active Comparator): ~90-second video of depressed cis-gender male
  Interventions: Behavioral: Short videos
- Transgender female (TF) (Active Comparator): ~90-second video of depressed transgender female
  Interventions: Behavioral: Short videos
- Cis-gender female (CF) (Active Comparator): ~90-second video of depressed cis-gender female
  Interventions: Behavioral: Short videos

INTERVENTIONS:
Behavioral: Short videos — Intervention videos will each be of 90-second duration and feature four underage professionals (ages 16) acting as simulated patients. All videos will focus on an empowered presenter with depression sharing their personal story regarding depression and describe how social supports from family, friends, and community, as well as professional help assisted them in overcoming symptoms of their illness. The actors will include a transgender male, a cis-gender male, a transgender female, and a cis-gender female.

SUMMARY:
The purposes of this new study are to test among adolescent viewers the utility of brief video-based interventions to:

1. reduce transphobia;
2. reduce depression-related stigma and increase likelihood of treatment-seeking; and
3. examine the role of viewer's sex (male / female / non-binary), race (Black vs non-Black), and sexual orientation (straight vs LGBQ) as independent factors on the outcomes of interest.

DETAILED DESCRIPTION:
Intervention videos will each be of ~100-second duration and feature four underage professionals (ages 16) acting as simulated patients. All videos will focus on an empowered presenter with depression sharing their personal story regarding depression. They will describe how social supports from family, friends, and community, as well as professional help assisted them in overcoming symptoms of the illness, as well as how being transgender may have had an impact on it. The four actors will include two males (one trans, one cis) and tow females (one trans, one cis).

Assessments will occur at baseline and post-intervention, and will include:

1. Demographics (baseline only);
2. Primary outcome:

   a. Attitudes toward Transgender Men and Women (ATTMW) scale.
3. Secondary outcome:

   1. Transgender attitudes: feelings thermometer, modeled after Norton et al 2013.
   2. Depression-related stigma (Depression Stigma Scale [DSS]);and
   3. Help-seeking (General Help-Seeking Questionnaire [GHSQ]).

For each of study we intend to randomly assign ~1,000 individuals aged 14-18 as follows:

Randomized, in equal proportions, and stratified by sex and race, to view one of four ~100-second videos:

1. Transgender male;
2. Cis-gender male);
3. Transgender female;
4. Cis-gender female.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Living in the US
* Ages 14 - 18

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Attitudes toward Transgender Men and Women (ATTMW) scale | Before / after viewing videos (within 10 minutes)
  Attitudes toward Transgender Men and Women (ATTMW; Billard, 2018) is a scale to measure transphobic attitudes. It is a 24-item scale consisting of two similar but non-identical 12-item subscales, one for transgender males (ATTM), and one for women (ATTW). In this study, the study team will assign only one of the two subscales, according to the condition that subjects as randomly assigned to: those viewing the transgender adolescent male will be assigned to the ATTM; those to the female, to the ATTW. The results of both subscales are compatible with each other and can be merged into a single ATMW score. Each of the items is a statement on which participants are asked to rate their agreement on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
  The first 9 items are the same for the ATTM and AATW. Items 10-12 are unique for each of the two scales. These

SECONDARY OUTCOMES:
Change in transgender attitudes: feelings thermometer | Before / after viewing videos (within 10 minutes)
  This study will utilize a scale called feelings thermometer, modeled after Norton and Herek, 2013:
  "Using a scale from zero to 100, please tell us your personal feelings toward each of the following groups of friends, teachers, or colleagues. As you do this task, think of an imaginary thermometer. The warmer or more favorable you feel toward the group, the higher the number you should give it. The colder or less favorable you feel, the lower the number. If you feel neither warm nor cold toward the group, rate it 50." To familiarize respondents with the response format, they will be first presented with thermometers for "Men in general" and "Women in general," with each respondent rating her or his own sex first. Next, they rate different gender groups (transgender males, transgender females). Higher ratings (maximum 100) indicate warmer, more favorable feelings toward the target whereas lower ratings (minimum 0) indicate colder, more negative feelings.
Change in Depression-related stigma (Depression Stigma Scale [DSS]; Personal component only): TOTAL SCORE | Before / after viewing videos (within 10 minutes)
  The DSS (Christensen, Jorm, Evans, & Groves, 2004) is a self-report instrument composed of two 9-item subscales. The first subscale measures the participants' own/ personal attitudes, and the second measures participants' beliefs about the attitudes of others ('Depression is sign of weakness' vs. 'Most people believe that depression is a sign of weakness'). The Personal subscale (DSS-Personal) will be used in this study. The DSS has a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). The total score comprises the sum of its item scores, and a higher score indicates more stigma (worse outcome). The DSS-Personal subscale has shown adequate psychometric properties: 0.71 test-retest reliability, 0.76 internal consistency (Griffiths et al., 2004). In our earlier study (Amsalem and Martin, 2021), Cronbach's a was .83.
Change in Help-seeking (General Help-Seeking Questionnaire [GHSQ]; Emotional and Suicide components): MEAN SCORE | Before / after viewing videos (within 10 minutes)
  The General Help-Seeking Questionnaire (GHSQ) (Wilson, Deane, Marshall, & Dalley, 2008) was developed to measure help-seeking intentions from different sources (friend, parent, mental health professional, and others) and is divided into personal-emotional problems and suicidal thoughts (Ibrahim et al., 2019). The instrument consists of 10 items for each part, each rated on a 0 (extremely unlikely) to 7 (extremely likely)Likert scale. Higher scores on this scale indicate more help seeking (better outcome).
  General stem:
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
Change in DSS Item 1 | Before / after viewing videos (within 10 minutes)
  DDS Item #1: People with depression could snap out of it if they wanted.
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5)
Change in DSS Item 2 | Before / after viewing videos (within 10 minutes)
  DDS Item #2: Depression is a sign of personal weakness
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 3 | Before / after viewing videos (within 10 minutes)
  DDS Item #3: Depression is not a real medical illness
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 4 | Before / after viewing videos (within 10 minutes)
  DDS Item #4: People with depression are dangerous
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 5 | Before / after viewing videos (within 10 minutes)
  DDS Item #5: It is best to avoid people with depression, so you don't become depressed yourself
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 6 | Before / after viewing videos (within 10 minutes)
  DDS Item #6: People with depression are unpredictable
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 7 | Before / after viewing videos (within 10 minutes)
  DDS Item #7: If I had depression, I would not tell anyone
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 8 | Before / after viewing videos (within 10 minutes)
  DDS Item #8 : I would not employ someone if I knew they had been depressed
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 9 | Before / after viewing videos (within 10 minutes)
  DDS Item #9: I would not vote for a politician if I knew they had been depressed
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in GHSQ Emotional Item 1 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Intimate partner (e.g., girlfriend, boyfriend)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 2 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Friend (not related to you)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 3 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Parent
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 4 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Other relative/family member
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 5 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Mental health professional (e.g., psychologist, social worker, counselor)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 6 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Phone helpline (e.g., lifeline)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 7 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Doctor/GP
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 8 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Minister or religious leader (e.g., Priest, Rabbi, Chaplain)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 9 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  I would not seek help from anyone
  **REVERSE SCORED ITEM** Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). LOWER scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 10 | Before / after viewing videos (within 10 minutes)
  If you were having a personal or emotional problem, how likely is it that you would seek help from the following people?
  Emotional Item # 10: I would seek help from another not listed above
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 1 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Intimate partner (e.g., girlfriend, boyfriend)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 2 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Friend (not related to you)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 3 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Parent
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 4 | Before / after viewing videos (within 10 minutes)
  Other relative/family member
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 5 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Mental health professional (e.g., psychologist, social worker, counselor)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 6 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Phone helpline (e.g., lifeline)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 7 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Doctor/GP
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 8 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  Minister or religious leader (e.g., Priest, Rabbi, Chaplain)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 9 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  GHSQ Item# 9: I would not seek help from anyone
  **REVERSE SCORED ITEM** Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). LOWER scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 10 | Before / after viewing videos (within 10 minutes)
  If you were having suicidal thoughts, how likely is it that you would seek help from the following people?
  GHSQ Item# 10:I would seek help from another not listed above
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in ATTMW Item 1 | Before / after viewing videos (within 10 minutes)
  ATTMW Item#1: Transgender men/women will never really be men/women
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 2 | Before / after viewing videos (within 10 minutes)
  ATTMW Item#2:Transgender men/women are not really men/women
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 3 | Before / after viewing videos (within 10 minutes)
  ATTMW Item#3:Transgender men/women are only able to look like men/women, but not be men/women
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 4 | Before / after viewing videos (within 10 minutes)
  ATTMW Item#4:Transgender men/women are unable to accept who they really are
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 5 | Before / after viewing videos (within 10 minutes)
  ATTMW Item#5:Transgender men/women are trying to be someone they're not
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 6 | Before / after viewing videos (within 10 minutes)
  Transgender adolescent men/women are denying their DNA
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 7 | Before / after viewing videos (within 10 minutes)
  ATTMW Item #8:Transgender men/women cannot just "identify" as men/women
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in **ATTM** Item 11 | Before / after viewing videos (within 10 minutes)
  ATTM Item #11: Transgender men are misguided
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 8 | Before / after viewing videos (within 10 minutes)
  ATTMW Item #10:Transgender men/women are unnatural
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in ATTMW Item 9 | Before / after viewing videos (within 10 minutes)
  ATTMW Item #11:Transgender men/women don't really understand what it means to be a man/woman
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in **ATTM** Item 11 | Before / after viewing videos (within 10 minutes)
  ATTMW Item #11:Transgender men are emotionally unstable
  Score on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in **ATTW** Item 11 | Before / after viewing videos (within 10 minutes)
  Transgender women are defying their nature.
Change in **ATTM** Item 10 | Before / after viewing videos (within 10 minutes)
  Transgender men seem absolutely normal to me (R)
  (R) = REVERSE-SCORED
  Scored on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in **ATTW** Item 10 | Before / after viewing videos (within 10 minutes)
  Transgender women only think they are females
  Scored on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.
Change in **ATTW** Item 12 | Before / after viewing videos (within 10 minutes)
  There is something unique about being a woman that transgender adolescent females can never experience
  Scored on a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater anti-transgender prejudice, while lower scores indicate less prejudice.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale Child Center, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths KM, Christensen H, Jorm AF, Evans K, Groves C. Effect of web-based depression literacy and cognitive-behavioural therapy interventions on stigmatising attitudes to depression: randomised controlled trial. Br J Psychiatry. 2004 Oct;185:342-9. doi: 10.1192/bjp.185.4.342. PMID 15458995
- [Background] Wilson CJ, Deane FP, Marshall KL, Dalley A. Adolescents' suicidal thinking and reluctance to consult general medical practitioners. J Youth Adolesc. 2010 Apr;39(4):343-56. doi: 10.1007/s10964-009-9436-6. Epub 2009 Jul 15. PMID 20229227
- [Background] Norton AT, Herek GM. Heterosexuals' attitudes toward transgender people: findings from a national probability sample of US Adults. Sex Roles. 2013;68(11-12):738-753. doi:10.1007/s11199-011-0110-6
- [Background] Billard TJ. Attitudes Toward Transgender Men and Women: Development and Validation of a New Measure. Front Psychol. 2018 Apr 3;9:387. doi: 10.3389/fpsyg.2018.00387. eCollection 2018. PMID 29666595
- [Derived] Amsalem D, Halloran J, Penque B, Celentano J, Martin A. Effect of a Brief Social Contact Video on Transphobia and Depression-Related Stigma Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220376. doi: 10.1001/jamanetworkopen.2022.0376. PMID 35212749